CLINICAL TRIAL: NCT05719948
Title: Combined Continuous and Pulsed Radiofrequency Ablation for Pain Relief and Their Safety in Cervical Facet Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Associate professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R 333
Record Dates: First submitted 2022-11-24; First posted 2023-02-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Radiofrequency Ablation
Keywords: medial branch; Neck pain; Radiofrequency ablation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: One model recieved continous RF while the other recieved combined pulsed and continous RF.
Who Masked: Investigator, Outcomes Assessor
Masking Description: None of the investigator or outcomees assessor know the intervention used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flouroscopic guidance cervical medial branch continous RF ablation (Active Comparator): After the patient lying prone we obtaining the posterior approach with PA view then lateral 15 degrees the C shaped edge of the cervical vertebrae were appeared and then we advance the needle till reaching this C shaped till hitting the bone then slipping the active tip slightly therafter we obtaining lateral view to determine the depth of the needle over the cervical pedicle.
  patients in the continous radiofrequency group will be underwent continous radiofrequency at 80°C for 90 seconds for 2 cycles
  Interventions: Procedure: Flouroscopic guidance cervical medial branch radiofrequency ablation
- Flouroscopic guidance cervical medial branch combined pulsed and continous RF ablation (Active Comparator): After the patient lying prone we obtaining the posterior approach with PA view then lateral 15 degrees the C shaped edge of the cervical vertebrae were appeared and then we advance the needle till reaching this C shaped till hitting the bone then slipping the active tip slightly therafter we obtaining lateral view to determine the depth of the needle over the cervical pedicle.
  patients in the continous and pulsed group will be underwent continous and pulsed radiofrequency at 80°C for 90 seconds for 1 cycle followed by pulsed radiofrequency at 42°C for 120 seconds for 1 cycle
  Interventions: Procedure: Flouroscopic guidance cervical medial branch radiofrequency ablation

INTERVENTIONS:
Procedure: Flouroscopic guidance cervical medial branch radiofrequency ablation — Electromagnetic wave deposition near nerve tissue for pain management

SUMMARY:
Continuous radiofrequency ablation (CRF) is the effective management for cervical facet joint pain but related with neuropathic symptoms in post-radiofrequency period. Additionally, pulse radiofrequency ablation (PRF) provides relief of neuropathic symptoms. However, the effect of CRF followed by PRF has yet to be validated

DETAILED DESCRIPTION:
Diagnostic procedure symptomatic facet joint was designated according to pain referral. Also, medial branches were injected with 2% lidocaine 0.3 ml per site.

Treatment procedure The posterior technique was first described in 1995 . All interventions assessed the intravenous saline lock on arrival at the outpatient department using pulse oximetry and noninvasive blood pressure monitoring and intravenous sedation as required. Patients were assigned in a prone position under C-ARM fluoroscopic guidance with a Neurotherm NT 2000 Lesion Generator the (USA manufactured) . The electrode pad of the radiofrequency equipment was attached to the ipsilateral side of the posterior thigh. After the skin was then anesthetized with 1% lidocaine, a 20-gauge, 10-cm cannula with 10-mm curved active tip (Diros RF Cannula, Diros Technology Inc., Canada) was inserted along a 15 to 30 degree angle to the sagittal plane (slightly posterior oblique approach) . The cannula was applied until reaching the lateral part of the articular pillar . Then the depth of the cannula was checked using a lateral view. A probe was inserted through the cannula and linked to a radiofrequency generator (Diros Technology OWL, Canada). After impedance were accomplished at below 500 Ohm, sensory stimulation was performed at 50 Hz and the patient reported not feeling any tingling sensation along the distribution of dermatome. Consequently, a motor stimulation (2 Hz) was executed until multifidus twitching was presented at stimulation less than 1 volts and no motor twitching was observed along the myotome. A non-ionic contrast medium was injected to ensure the intravascular injection before 1% lidocaine 0.5 ml was injected after the needle reached the desired location. The study investigated two lesions due to the anatomical variation of the medial branches. Patients in the CRF group (n = 16) underwent CRF at 80°C for 90 seconds for 2 cycles. Patients in the CPRF group underwent CRF at 80°C for 90 seconds for 1 cycle followed by PRF at 42°C for 120 seconds for 1 cycle. 0.125% bupivacaine plus 2 mg of dexamethasone in a total volume of 1 mL were injected after lesioning had performed.

Measurement The demographic data including age, sex, comorbidities, body mass index (BMI), level of procedure, visual analog scale (VAS;1-100) Neck Pain Disability Index and complications were reviewed. It contains ten sectors: seven sectors related to everyday existing behaviors, two sectors correlated to pain, and one sector correlated to concentration. All items are marked from 0 to 5. A mark of 0 denotes the maximum level of function, while a mark of 5 indicates the bottom level of function. The maximum mark is 50, and a greater mark relates to an increased level of disability. The NDI scores were recorded before intervention and first month, third month, sixth month, ninth months and 12 months after intervention. The follow-up was performed either face to face or by phone, and patients were not permitted to use over-the counter analgesic medication. The primary outcome was number of patients who had successful treatment, expressed as at least 80% pain relief from baseline and NDI score less than 15 for at least 3 months . The secondary outcomes comprised the duration of pain relief defined as the time of pain relief until VAS had restored to at least 50% from baseline and side effects including numbness, ataxia, dysesthesia, hypersensitivity, itching and muscular weakness (dropped head syndrome) between group comparisons. A research assistant, who was uninvolved in the intervention or post-operative follow-up, collected all data in prospective medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients age from (30-75) years old.
* ASA ( I, II).
* Patients presenting positive diagnostic cervical medial branche block defined as pain relief more than 50% from baseline.

Exclusion Criteria:

* Repeated cervical radiofrequency ablation.
* Patients presenting neck pain with radicular symptoms.
* Previous cervical discectomy or fixation surgery.
* Malignancy.
* local infection
* Psychological problem.
* language barrier.
* History of allergy to radio-opaque contrast solution,lidocaine or bupivacaine. - Inadequate medical proplem (hepatic, renal, cardiac) patients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
neck disability index pre and post-intervention between comparison groups | One month
  Neck disability index : It contains ten sectors: seven sectors related to everyday existing behaviors, two sectors correlated to pain, and one sector correlated to concentration. All items are marked from 0 to 5. A mark of 0 denotes the maximum level of function, while a mark of 5 indicates the bottom level of function. The maximum mark is 50, and a greater mark relates to an increased level of disability.
neck disability index pre and post-intervention between comparison groups | 3 months
  Neck disability index : It contains ten sectors: seven sectors related to everyday existing behaviors, two sectors correlated to pain, and one sector correlated to concentration. All items are marked from 0 to 5. A mark of 0 denotes the maximum level of function, while a mark of 5 indicates the bottom level of function. The maximum mark is 50, and a greater mark relates to an increased level of disability.
neck disability index pre and post-intervention between comparison groups | 6 months
  Neck disability index : It contains ten sectors: seven sectors related to everyday existing behaviors, two sectors correlated to pain, and one sector correlated to concentration. All items are marked from 0 to 5. A mark of 0 denotes the maximum level of function, while a mark of 5 indicates the bottom level of function. The maximum mark is 50, and a greater mark relates to an increased level of disability.
neck disability index pre and post-intervention between comparison groups | 12 months
  Neck disability index : It contains ten sectors: seven sectors related to everyday existing behaviors, two sectors correlated to pain, and one sector correlated to concentration. All items are marked from 0 to 5. A mark of 0 denotes the maximum level of function, while a mark of 5 indicates the bottom level of function. The maximum mark is 50, and a greater mark relates to an increased level of disability.
VAS SCORE | One month
  of procedure, visual analog scale (VAS;1-100)
VAS SCORE | 3 months
  of procedure, visual analog scale (VAS;1-100)
VAS SCORE | 6 months
  of procedure, visual analog scale (VAS;1-100)
VAS SCORE | 12 months
  of procedure, visual analog scale (VAS;1-100)

SECONDARY OUTCOMES:
Duration of pain relief | One month, 3months,6 months, 12 months
  The duration of pain relief was expressed as the period between pain relief and pain reoccurrence to 50% of pre-procedural pain level
Complications | One month, 3 months, 6months, 12 months
  Numbness, dysethesia, drop head syndrome, hypersensitivity, ataxia

CONTACTS AND LOCATIONS:
Locations (1):
- Atef Mohamed mahmoud, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be given on resonable request